CLINICAL TRIAL: NCT00370305
Title: The Pathogenic Role of 11ß-hydroxysteroid Dehydrogenase in the Metabolic Syndrome - the Effect of Rosiglitazone
Brief Title: 11ß-HSD1 and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Professor Joachim Spranger, Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ek. 211-02d
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Syndrome; Impaired Glucose Tolerance
Keywords: 11ß-hydroxysteroid dehydrogenase; rosiglitazone; insulin sensitivity; Impaired glucose tolerance
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Insulin Resistance | interventions — Rosiglitazone

ARMS (1):
- Rosiglitazone treatment (Experimental): Rosiglitazone will be given to the subjects. All subjects will be analyzed before and after treatment
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — 89 mg BID for 8 weeks, orally
  Other Names: Avandia

SUMMARY:
The purpose of this study is to determine whether the insulin sensitizing effects of rosiglitazone were accompanied by changes in 11ß-HSD1 expression and activity in different tissues. Furthermore the metabolic and hormonal effects of PPAR gamma stimulation by rosiglitazone will be analysed in several tissues.

DETAILED DESCRIPTION:
The PPARgamma agonist rosiglitazone (R) increases insulin sensitivity, which is comparable to the effects of a reduction in 11ß-hydroxysteroid dehydrogenase type 1 (11β-HSD1) activity in animal models. We therefore aimed to investigate whether rosiglitazone-induced insulin sensitivity is associated with changes in 11β-HSD1 activity in different tissues in subjects suffering from impaired glucose tolerance. Furthermore the metabolic and hormonal effects of PPAR gamma stimulation by rosiglitazone will be analysed in those tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance

Exclusion Criteria:

* Treatment with insulin
* Orally taken antidiabetic medication, glucocorticoids or vitamin K-antagonists
* Heart failure
* Impaired hepatic or renal function
* Anaemia
* Disturbed coagulation
* Any other endocrine disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
changes of 11ß-HSD1 expression in adipose tissue and skeletal muscle during 8 weeks of rosiglitazone treatment | 8 weeks
  11ß-HSD1 expression will be measured in adipose tissue and skeletal muscle
changes of hepatic 11ß-HSD1 activity during 8 weeks of rosiglitazone treatment | 8 weeks
  11ß-HSD1 activity will be assessed by measuring conversion of cortisone to cortisol (ratio will be calculated)
changes of whole body 11ß-HSD1 activity during 8 weeks of rosiglitazone treatment | 8 weeks
  whole body 11ß-HSD1 activity will be assessed by measuring the ratio of urinary tetrahydrocortisol (THF) + alpha-tetrahydrocortisol (THF) / tetrahydrocortisone

SECONDARY OUTCOMES:
changes in insulin sensitivity during 8 weeks of rosiglitazone treatment | 8 weeks
  Measurement of whole body and myocellular insulin sensitivity (mg•kg-1•min-1/(mU•L-1)) before and after treatment
Hormonal and metabolic changes induced by the intervention | 3 months
  Whole body as well as tissue specific (skeletal muscle and different adipose tissue compartment) changes in hormonal circuits and metabolism will be analyzed
changes of FGF-21 induced by the intervention | 8 weeks
  FGF-21 (ng/ml) will be assessed in plasma samples
changes of free fatty acids (FFA) induced by the intervention | 8 weeks
  FFA (mmol/l) will be assessed in plasma samples
changes of myocellular SCD1 expression induced by the intervention | 8 weeks
  myocellular SCD1 mRNA expression will be assessed
changes of myocellular long chain fatty acids (LC-FA) expression induced by the intervention | 8 weeks
  myocellular LC-FA mRNA expression will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Knut Mai, Principal Investigator — Charite, Dpt. of Endocrinology, Diabetes and Nutrition
Locations (1):
- Charite, Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Mai K, Andres J, Bobbert T, Assmann A, Biedasek K, Diederich S, Graham I, Larson TR, Pfeiffer AF, Spranger J. Rosiglitazone increases fatty acid Delta9-desaturation and decreases elongase activity index in human skeletal muscle in vivo. Metabolism. 2012 Jan;61(1):108-16. doi: 10.1016/j.metabol.2011.05.018. Epub 2011 Jul 7. PMID 21741058